CLINICAL TRIAL: NCT06018753
Title: Umbrella Study for Analysis of Data Related to Patients With Cancer
Acronym: Polaris
Status: Recruiting | Type: Observational
Sponsor: Tempus AI (Industry)
Responsible Party: Sponsor
Other Study IDs: TP-CA-005; Pro00073040 (Other: Advarra)
Record Dates: First submitted 2023-08-15; First posted 2023-08-31 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Cancer
Keywords: Data Analysis; Master Protocol; Oncology; Retrospective
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with cancer: No intervention or sample collection is required on the study.

SUMMARY:
This study is a multisite, minimal risk, non-interventional study using patient electronic health record data collected as part of standard of care to answer cohort-based research questions and create robust real-world data sets.

DETAILED DESCRIPTION:
One key purpose of the Study is to collect data that may be used for a wide range of scientific questions and real-world insights.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be diagnosed with cancer
* Medical records available to meet cohort requirements

Exclusion Criteria:

- None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population of subjects targeted are: 1) those who have cancer, and 2) those for whom medical records are available.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Provide RWD/E Datasets to Research Collaborators to Support Development | 5 years
  Use data analysis to enable deeper understanding of patient population characteristics and outcomes to more accurately assess clinical trial feasibility and optimize trial design.
Provide RWD/E Datasets to Research Collaborators to Support Regulatory | 5 years
  Use data analysis to generate supplemental data for new accelerated approval pathway filings and provide real world control arms where necessary.
Provide RWD/E Datasets to Research Collaborators to Support Commercialization | 5 years
  Use data analysis to enable more precise characterization of biomarker testing rates, factors influencing access to testing, and uptake of recently approved therapies to inform commercial strategy for pharmaceutical companies and generate evidence for payors.
Provide RWD/E Datasets to Research Collaborators to Support Phase IV Surveillance | 5 years
  Use data analysis to support post approval understanding of longer term side effects that may not be sufficiently detected via randomized clinical trials.
Provide RWD/E Datasets to Research Collaborators to Support Real-World Insights | 5 years
  Use data analysis to further understanding of variations in patient care across the US to help ensure patients have access to optimal testing and treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Rhodes, MD, Study Director — Tempus AI, Inc.
Locations (10):
- United States (10):
  - Memorial Health Services, Fountain Valley, California
  - Cancer Specialists of Northern Florida, Jacksonville, Florida
  - Hawaii Cancer Care, Honolulu, Hawaii
  - Illinois Cancer Care, Peoria, Illinois
  - Northwest Oncology and Hematology, Rolling Meadows, Illinois
  - Community Health Network, Indianapolis, Indiana
  - Southcoast Centers for Cancer Care, Fairhaven, Massachusetts
  - Sanford Fargo, Fargo, North Dakota
  - Taylor Cancer Research Center, Maumee, Ohio
  - Avera Cancer Institute, Sioux Falls, South Dakota

REFERENCES:
- [Background] Thomas M. Pharma and the benefits of Real World Data. Drug Discovery World (DDW). Published November 4, 2021. Accessed May 5, 2023. https://www.ddw-online.com/trends-analysis-pharma-and-the-benefits-of-real-world-data-13702-202111/
- [Background] Office of the Commissioner. Oncology Real World Evidence Program. U.S. Food and Drug Administration. Accessed May 5, 2023. https://www.fda.gov/about-fda/oncology-center-excellence/oncology-real-world-evidence-program
- [Background] Grayson N. Real-world data can help make better drugs and do it faster. STAT. Published May 2, 2018. Accessed May 5, 2023. https://www.statnews.com/2018/05/02/real-world-data-drug-development/
- [Background] Rudrapatna VA, Butte AJ. Opportunities and challenges in using real-world data for health care. J Clin Invest. 2020 Feb 3;130(2):565-574. doi: 10.1172/JCI129197. PMID 32011317